CLINICAL TRIAL: NCT04890470
Title: Effects of Oxytocin and Vasopressin on Moral Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-78
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: moral decision making; oxytocin; vasopressin
MeSH Terms: conditions — Diabetes Insipidus | interventions — Oxytocin; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oxytocin group (Experimental): subjects with oxytocin treatment
  Interventions: Drug: Oxytocin
- vasopressin group (Experimental): subjects with vasopressin treatment
  Interventions: Drug: Vasopressin
- placebo group (Placebo Comparator): subjects with placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — intranasal administration of oxytocin (24 IU)
  Arms: oxytocin group
Drug: Vasopressin — intranasal administration of vasopressin (20 IU)
  Arms: vasopressin group
Drug: Placebo — intranasal administration of placebo
  Arms: placebo group

SUMMARY:
To determine whether the neuropeptide oxytocin (OXT) and vassopressin (AVP) influence moral decision making

DETAILED DESCRIPTION:
In a double-blind, between- subject placebo (PLC) controlled design, subjects will first complete a series of questionnaires in terms of mood, clinical symptoms, and traits. After that their moral judgment and emotion towards both verbal descriptions of moral dilemma scenarios and pictures of specific interpersonal ones will be assessed and the effect of intranasal OXT and AVP between both male and female healthy subjects will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Effect of OXT and AVP on behavioral index of moral decision task | 45 mins - 105 mins
  intensity of feelings

CONTACTS AND LOCATIONS:
Overall Officials: Keith M. Kendrick, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- Xiaoxiao Zheng, Sichuan, Sichuan, China